CLINICAL TRIAL: NCT03981432
Title: Identification of the Physical and Dietary Profile on Constitutionally Lean People: the NUTRILEAN Study
Brief Title: Energy Intake, Exercise and Constitutional Leanness
Acronym: Nutrilean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2018 DUCLOS 3
Record Dates: First submitted 2019-04-29; First posted 2019-06-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Anorexia Nervosa; Constitutional Leanness
Keywords: appetite control; leanness; physical fitness
MeSH Terms: conditions — Anorexia Nervosa; Thinness

STUDY DESIGN:
Intervention Model Description: all participants receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Constitutional leanness (Experimental): Constitutional leanness
  Interventions: Behavioral: REST-Fixed; Behavioral: REST-AdLib; Behavioral: EX-AdLib
- Normal weight (Experimental): Normal weight women
  Interventions: Behavioral: REST-Fixed; Behavioral: REST-AdLib; Behavioral: EX-AdLib
- Anorexia nevrosa (Experimental): women presenting Anorexia nevrosa
  Interventions: Behavioral: REST-Fixed; Behavioral: REST-AdLib; Behavioral: EX-AdLib

INTERVENTIONS:
Behavioral: REST-Fixed — condition without exercise / rest condition. The participants will be asked to remain quiet and at rest during the morning and will receive a fixed meal at lunch. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
Behavioral: REST-AdLib — condition without exercise / rest condition. The participants will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at lunch. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
Behavioral: EX-AdLib — condition with an acute exercise set 30 minutes before the lunch meal that will be served ad libitum This will be a 30-minute exercise set at 65% of their capacities (cycling), 30 minutes before lunch.

SUMMARY:
The aim of this study will be to identify the physical and dietary profile of adult women presenting constitutional leanness (CL), comparatively with normal-weight peers and BMI-matched women with anorexia nervosa. After an evaluation of their daily energy intake, physical activity level, body composition, aerobic capacities and muscle strength, women from the normal weight and CL groups will be asked to realized laboratory sessions to evaluate their energy intake and appetite feelings responses to acute exercise

DETAILED DESCRIPTION:
Body composition (using X-ray absorptiometry), muscle strength (biodex), daily energy intake (dietary record), food preferences (Leeds Food Preference Questionnaire) and physical activity level (GT3X accelerometers) will be assessed among women with constitutional leanness normal weight women and women with anorexia nervosa. The CT and NW groups will then be asked to randomly realized three experimental session: i) a rest session with an fixed lunch meal; a rest session with an ad libitum meal ; iii) an exercise session with an ad libitum meal. Their ad libitum energy intake will be assessed during the two last sessions. Appetite feelings will be assessed at regular intervals and their food reward in response to the lunch will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Common criteria to the three groups
* Women
* Aged 18 to 35 years old

  -- Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Criteria specific to constitutionally lean women

* BMI ≤ 17.5 kg/m2
* Weight stable for the last three months
* No dietary disorders
* no sign of denutrition
* absence of amenorrhea

Criteria specific to women with anorexia nervosa

* BMI ≤ 17.5 kg/m2
* Pure restrictive Anorxia nevrosa: no binge eating or vomiting episodes for the last thress months.
* DSM V (2013) crietria Criteria specific to normal weight women
* 20 kg/m2 ≤ BMI ≤ 25 kg/m2
* Weight stable for the last three months
* No dietary disorders
* no sign of denutrition
* absence of amenorrhea

Exclusion Criteria:

* Pregnancy
* Intensive physical activity level (aboce 3 sessions per week)
* Impaired level of IGF-1, estradiol, T3free, cortisol and leptin (for normal weight and constitutionally lean women)
* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* Medication that could interfer with the study.
* cardiovascular disease or risks
* Surgery within the last 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change in energy intake measured during the ad libitum buffet meal (in kcal). | day 1 , day 8
  food intake will be measured ad libitum during a lunch buffet. The participants will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software.

SECONDARY OUTCOMES:
Body fat mass | day 1
  the percentage of body fat and the quantity of fat mass will be assessed using X-ray absorptiometry (DXA)
fat free mass | day 1
  the percentage of body fat and the quantity of fat mass will be assessed using X-ray absorptiometry (DXA)
Physical activity level | day 1
  The time spent at low-moderate and vigorous physical activity will be assessed using a 7-day accelerometry record (Actigraph GT3X)
Daily energy intake | Trough 3 days
  The amount and quality of food intake will be assessed using a three-day dietary record
Food reward | day 1 , day 8 , day 15
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ)
change in energy intake measured during the ad libitum buffet meal (in kcal). | day 1 , day 8
  food intake will be measured ad libitum during a lunch buffet. The participants will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software
Hunger feelings | day 1 , day 8 , day 15
  hunger area under the curve will be assessed using visual analogue scale through a the day using a visual analog scale from 0 millimeter (no sensation) to 100mm (highest sensation)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France